CLINICAL TRIAL: NCT04194996
Title: Prospective Radiographic and Clinical Evaluation of Surgical Treatment for Cervical Deformity: A Multi-Center Study 2.0
Brief Title: Radiographic and Clinical Evaluation of Surgical Treatment for Cervical Deformity: A Multi-Center Study 2.0
Acronym: PCD 2
Status: Recruiting | Type: Observational
Sponsor: International Spine Study Group Foundation (Other)
Collaborators: DePuy Synthes (Industry); Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2131
Record Dates: First submitted 2019-11-25; First posted 2019-12-11 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Cervical Deformity
Keywords: Cervical deformity; Kyphosis; Scoliosis
MeSH Terms: conditions — Kyphosis; Scoliosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Operative: Inclusion criteria:
  1. ≥18 years old at time of treatment
  2. Diagnosis of cervical deformity- must meet one or more of the following criteria:
     * C2-C7 sagittal kyphosis (Cobb > 15o)
     * T1S-CL > 35o
     * Segmental cervical kyphosis > 10o between any 2 vertebra between C2-T1 or > 15o across any 3 vertebra between C2-T1
     * Cervical scoliosis > 10o (Cobb angle must include end vertebra within the cervical spine)
     * C2-C7 SVA > 4cm
     * McGregor's slope > 20 degrees or CBVA > 25 degrees
  3. Plan for surgical correction of cervical deformity in the next 6 months
  Interventions: Procedure: Surgical intervention

INTERVENTIONS:
Procedure: Surgical intervention — Surgical interventions will be patient specified by treating surgeon.

SUMMARY:
Multi-center, prospective, non-randomized study to evaluate outcomes of surgically treated patients with adult cervical spinal deformity.

DETAILED DESCRIPTION:
Adult cervical deformity (ACD) is an uncommon but potentially severely debilitating condition with a broad range of causes that include but are not limited to spondylosis, inflammatory arthropathy, trauma, infection, iatrogenic, neoplastic, congenital, and neuromuscular processes. In general, sagittal plane deformities typically produce kyphosis, and coronal plane deformities result in scoliosis. Cervical kyphotic deformities are most commonly encountered in the setting of prior surgical destabilization, while cervical scoliosis is most commonly associated with congenital and neuromuscular conditions.

Cervical kyphosis may be progressive and can result in neurological symptoms, including myelopathy. The most severe forms, such as those associated with spondylotic arthropathies, can produce "chin-on-chest" deformity, which can compromise horizontal gaze, swallowing, and breathing. Even in the absence of these conditions, cervical deformity is often associated with pain and functional disability. For adult thoracolumbar deformities, substantial efforts have been made to characterize clinical presentations, develop standardized classification systems, define optimal treatment approaches, describes operative complication rates, and to present structured clinical outcomes. However, despite the potential for profound impact of cervical deformity on function and health-related quality of life, there remains a remarkable paucity of high-quality studies that address these complex conditions.

Health professionals providing nonoperative and surgical care for these patients are left to make important treatment decisions based on a combination of personal experience, anecdotal experience of colleagues and experts, and relatively small, often single-surgeon or single-center, retrospective case reports or case series in the literature. Recent systematic reviews have high-lighted the lack of studies relevant to cervical deformity and have failed to identify any prospective studies.

The International Spine Study Group (ISSG) consists of orthopedic and neurological spine surgeons with a practice emphasis on spinal deformity patients. These surgeons, from 12 busy surgical centers, meet regularly to design and perform clinical research focused on spinal deformity, including successful prospective enrollment of more than 1,000 adult thoracolumbar deformity patients into the ISSG database. This group has a proven track record and regularly presents a substantial number of abstracts to the major spine meetings and has an extensive publication record.

The ISSG members have currently enrolled more than 150 patients into the first generation prospective cervical deformity database and have produced approximately 50 abstracts and more than 25 manuscripts to date with the resulting data. The group has learned extensively from this first-generation database, but there is much yet to learn, as the literature remains relatively sparse on the topic of adult cervical deformity. Based on what we have learned from the first generation database; we have substantially modified the inclusion criteria for this second generation database. In addition, several new outcomes measures and functional assessments will be collected at baseline and follow-up intervals as part of this current proposal.

The resources of the ISSG offer an unprecedented opportunity to create a prospectively collected multicenter database of cervical deformity patients that includes standardized health-related quality of life measures at baseline and regular follow-up, clinical and surgical parameters, and complications. The database and questionnaires have been carefully redesigned based on what we have learned in order to better collect data that will help to clarify many of the unresolved issues that are important for the care of cervical deformity patients. This project has substantial potential to significantly impact the field of cervical deformity and the care of deformity patients beyond what we have already been able to accomplish based on the first generation cervical deformity database. Herein we propose the second iteration for this project that promises to further advance our evolving understanding of these complex deformities.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old at time of treatment
* Diagnosis of cervical deformity- must meet one or more of the following criteria:

  * C2-C7 sagittal kyphosis (Cobb > 15 degrees)
  * T1S-CL > 35o
  * Segmental cervical kyphosis > 10 degrees between any 2 vertebra between C2-T1 or > 15 degrees across any 3 vertebra between C2-T1
  * Cervical scoliosis > 10 degrees (Cobb angle must include end vertebra within the cervical spine)
  * C2-C7 SVA > 4cm
  * McGregor's slope > 20 degrees or CBVA > 25 degrees
* Plan for surgical correction of cervical deformity in the next 6 months
* Willing to provide consent and complete study forms at baseline and follow-up intervals

Exclusion Criteria:

* Active spine tumor or infection
* Deformity due to acute trauma
* Unwilling to provide consent or to complete study forms
* Prisoner
* Pregnant or immediate plans to get pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spine Surgeon Clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2033-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain Numeric rating scale (NRS) - Headaches | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Self-reported pain in Head where 0=no pain/10=severe pain
Pain Numeric rating scale (NRS) - Neck | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Self-reported pain in Neck where 0=no pain/10=severe pain
Pain Numeric rating scale (NRS) - Upper extremity | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Self-reported pain in Arms where 0=no pain/10=severe pain
Pain Numeric rating scale (NRS) - Lower extremity | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Self-reported pain in Legs where 0=no pain/10=severe pain
Pain Numeric rating scale (NRS) - Back | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Self-reported pain in Back where 0=no pain/10=severe pain
Neck Disability Index (NDI) | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Patient reported neck disability tool
Veterans RAND 12 Item Health Survey (VR-12) | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Anxiety | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PROs
Patient-Reported Outcome Measurement Information System (PROMIS) - Depression | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PROs
Patient-Reported Outcome Measurement Information System (PROMIS) - Pain Interference | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PROs
Patient-Reported Outcome Measurement Information System (PROMIS) - Physical Function | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PROs
Patient-Reported Outcome Measurement Information System (PROMIS) - Social Satisfaction (Role) | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PROs
Patient-Reported Outcome Measurement Information System (PROMIS) - Social Satisfaction (DSA) | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PROs
Spine Radiographs | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Radiographic parameters (Cervical lordosis, Kyphosis, Scoliosis; Global balance in coronal and sagittal planes of the spine; pelvic parameters (pelvic incidence, tilt, slope) and bony fusion status.
Modified Japanese Orthopaedic Association Scale (mJOA) | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Patient reported outcome measuring functional status using scale of 0 to 18. The higher the score, the less disability.

SECONDARY OUTCOMES:
EAT-10 | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Measures swallowing difficulties as reported by the patient.
Voice Handicap Index (VHI-10) | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Measures voice handicap as reported by the patient.
Adverse evnts | 3 months and 1, 2, 5 & 10 year post treatment
  Any adverse events occurring & meeting study established reporting criteria
Edmonton Frail Scale | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Frailty scale from 0 to 17 where the higher the score the more frail the patient
CHSF Frail Scale | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  Clinical Frailty Scale from 1 to 9 where the higher the score, the more frail the patient
Dynamometer Hand Grip Strength test | Change from Preop to 3 months, 6 months and 1, 2, 5 & 10 year follow-up
  With patient seated, patient will squeeze dynamometer as hard as he/she can with each hand.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Smith, MD, Principal Investigator — University of Virginia, Department of Neurosurgery; Christopher Ames, MD, Principal Investigator — University of California, San Francisco, Department on Neurosurgery; Christopher I Shaffrey, MD, Principal Investigator — Duke University, Departments of Neurosurgery and Orthopaedic Surgery
Locations (17):
- United States (17):
  - Shiley Center for Orthopaedic Research and Education at Scripps Clinic, La Jolla, California
  - University of California Davis, Department of Orthopedic Surgery, Sacramento, California
  - University of California-San Francisco Medical Center, San Francisco, California
  - Denver International Spine Center, Rocky Mountain Hospital for Children and Presbyterian St. Luke's Medical Center, Denver, Colorado
  - Rush University, Department of Neurosurgery, Chicago, Illinois
  - University of Kansas Medical Center, Department of Orthopedic Surgery, Kansas City, Kansas
  - Leatherman Spine Center, Department of Orthopedic Surgery, Louisville, Kentucky
  - Johns Hopkins University, Department of Neurological Surgery, Baltimore, Maryland
  - University of Michigan, Department of Neurosurgery, Ann Arbor, Michigan
  - Washington University, Department of Orthopedic Surgery, St Louis, Missouri
  - Hospital for Special Surgery, Department of Orthopedic Surgery, New York, New York
  - New York University, Department of Orthopedic Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Health System, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical City Spine Hospital - Southwest Scoliosis Institute, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No